CLINICAL TRIAL: NCT07123376
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase I Clinical Study Was Conducted to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of HRS-9231 Injection in a Single Dose in Healthy Chinese Subjects
Brief Title: Pharmacokinetics, Pharmacodynamics Profile and Tolerance of HRS-9231 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Diagnostic
Other Study IDs: HRS-9231-101
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): 8 healthy subjects were to be included
  Interventions: Drug: HRS-9231; Drug: Placebo
- Group 2 (Experimental): 8 healthy subjects were to be included
  Interventions: Drug: HRS-9231; Drug: Placebo
- Group 3 (Experimental): 8 healthy subjects were to be included
  Interventions: Drug: HRS-9231; Drug: Placebo
- Group 4 (Experimental): 8 healthy subjects were to be included
  Interventions: Drug: HRS-9231; Drug: Placebo
- Group 5 (Experimental): 8 healthy subjects were to be included
  Interventions: Drug: HRS-9231; Drug: Placebo

INTERVENTIONS:
Drug: HRS-9231 — HRS-9231 was administered intravenously;
Drug: Placebo — Placebo was administered intravenously.

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic characteristics of HRS-9231 injection in a single dose in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 45 years.
2. Body mass index (BMI) of 19.0 to 28.0 kg/m2 (inclusive).
3. Understand in detail the content, procedure and possible adverse effects of the trial, and voluntarily sign the written informed consent form (ICF).

Exclusion Criteria:

1. Patients with contraindications for magnetic resonance imaging (MRI) examinations.
2. During the screening period, those whose 12-lead electrocardiogram examination is judged by clinical doctors as abnormal and of clinical significance will be selected.
3. Those with a history of drug abuse, drug use, or positive results in drug abuse screening.
4. Unable to tolerate venipunctures or have a history of fainting needles and blood.
5. People with various urinary disorders (such as frequent urination, difficulty in urination, etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Adverse events, serious adverse events | From ICF signing date to Day10

SECONDARY OUTCOMES:
Cmax：maximum concentration measured. Blood samples were taken to assess HRS-9231 concentration | From baseline (1 hour before injection) to 12 hours post-injection
t1/2 = terminal elimination half-life of the compound | From baseline (1 hour before injection) to 12 hours post-injection
Cl = total clearance | From baseline (1 hour before injection) to 12 hours post-injection

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided